CLINICAL TRIAL: NCT07099989
Title: A Randomized, Open-Label, 2-Cohort, 2-Period Crossover Study to Evaluate the Pharmacokinetics of GATE-251 (Zelquistinel), 3 and 10 mg, Under Both Fasted and Fed Conditions in Healthy Adult Participants
Brief Title: Pharmacokinetics of GATE-251 in Fasted or Fed State
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Syndeio Biosciences, Inc (Industry)
Collaborators: Dr. Vince Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GATE-251-C-110
Record Dates: First submitted 2025-07-21; First posted 2025-08-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers in Fed and Fasted State
Keywords: GATE-251; zelquistinel; N-methyl-D-aspartate (NMDA) receptor positive allosteric modulator; pharmacokinetics
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Zelquistinel, 3 mg Fasted (Active Comparator): Subjects will be randomized to one of two sequences. Subjects will be dosed with GATE-251, 3 mg oral tablet, during each sequence. Each subject will serve as their own control.
  Interventions: Drug: Zelquistinel 3 mg
- Zelquistinel, 3 mg Fed (Active Comparator): Subjects will be randomized to one of two sequences. Subjects will be dosed with GATE-251, 3 mg oral tablet, during each sequence. Each subject will serve as their own control.
  Interventions: Drug: Zelquistinel 3 mg
- Zelquisitinel, 10 mg Fasted (Active Comparator): Subjects will be randomized to one of two sequences. Subjects will be dosed with GATE-251, 10 mg oral tablet, during each sequence. Each subject will serve as their own control.
  Interventions: Drug: Zelquistinel 10 mg
- Zelquistinel, 10 Fed (Active Comparator): Subjects will be randomized to one of two sequences. Subjects will be dosed with GATE-251, 10 mg oral tablet, during each sequence. Each subject will serve as their own control.
  Interventions: Drug: Zelquistinel 10 mg

INTERVENTIONS:
Drug: Zelquistinel 3 mg — Subjects will receive Zelquistinel 3 mg in fed and fasted state (high fat meal).
  Arms: Zelquistinel, 3 mg Fasted; Zelquistinel, 3 mg Fed
Drug: Zelquistinel 10 mg — Subjects will receive Zelquistinel 10 mg in fed and fasted state (high fat meal).
  Arms: Zelquisitinel, 10 mg Fasted; Zelquistinel, 10 Fed

SUMMARY:
The primary purpose of this study is to assess the effect of food on the rate and extent of absorption of a single dose of GATE-251 3 mg or 10 mg oral tablets tablets in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a randomized, open-label, single-dose, 2-cohort, 2-period crossover study to assess the effect of food on the pharmacokinetics, safety, and tolerability of GATE-251 tablet in healthy adult participants. Two dose levels, 3 and 10 mg, will each be evaluated for food effect, 1 dose level per cohort, with approximately 32 participants (16 per cohort).

* Cohort 1: GATE-251, 3 mg single oral tablet administered under fasted and fed conditions
* Cohort 2: GATE-251, 10 mg single oral tablet administered under fasted and fed conditions

Study Design: This is a randomized, open-label, single-dose, 2-cohort, 2-period crossover study to assess the effect of food on the pharmacokinetics, safety, and tolerability of GATE-251 tablet in healthy adult participants. Two dose levels, 3 and 10 mg, will each be evaluated for food effect, 1 dose level per cohort, with approximately 32 participants (16 per cohort).

* Cohort 1: GATE-251, 3 mg single oral tablet administered under fasted and fed conditions
* Cohort 2: GATE-251, 10 mg single oral tablet administered under fasted and fed conditions After meeting eligibility requirements, participants will be admitted to the clinical research unit on Day -1. Participants within each cohort will be randomly assigned in a 1:1 ratio to a treatment sequence. Cohorts will be enrolled sequentially. Participants will only participate in 1 cohort.

On Day 1 of each period, participants will receive one of the following treatments:

* Treatment A (reference): GATE-251, 3 mg tablet, fasted conditions
* Treatment B (test): GATE-251, 3 mg tablet, fed conditions (high-fat, high-calorie meal)
* Treatment C (reference): GATE-251, 10 mg tablet, fasted conditions
* Treatment D (test): GATE-251, 10 mg tablet, fed conditions (high-fat, high-calorie meal) Fasted and fed conditions and test meal composition are defined by FDA guidance. For the fasted condition, GATE-251 will be administered after an overnight fast of at least 10 hours.

For the fed condition, after an overnight fast of at least 10 hours, participants will start the test meal approximately 30 minutes before administration of GATE-251. The test meal will be entirely consumed within 30 minutes.

For both fasted and fed conditions, GATE-251 will be administered with approximately 240 mL of water. Up to 200 mL of additional water will be allowed in increments of 50 mL, as needed. No water will be allowed for at least 1 hour before or after GATE-251 administration, except for the water consumed during administration. No food will be allowed for at least 4 hours after GATE-251 administration. In addition, participants will be semi-recumbent during the test meal and for at least 4 hours after study drug administration, except for when procedures or adverse events require the supine position.

The test meal will be a standard high-fat, high-calorie meal consisting of approximately 1000 calories with approximately 50% of the total calories from fat.

There will be a 7-day washout interval between doses then participants will cross over to Period 2 and receive GATE-251 at the same dose as in Period 1 under the alternate fasted or fed condition. Participants will be confined to the clinical study unit from Study Day -1 through Study Day 10 and will return on approximately Study Day 15 (7±2 days from the last dose) for the Follow-Up Visit (end of study).

Samples will be collected for pharmacokinetic analysis at the following timepoints for plasma, urine, and CSF.

* Plasma: On Day 1 of each period, blood samples will be collected at: 0 (pre-dose) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours after dosing.
* Urine: On Day 1 of each period, urine samples will be collected at: 0 (pre-dose) and 0-4-, 4-8-, 8-12-, and 12-24-hour intervals after dosing.
* Cerebrospinal fluid (CSF) collection: On Day 1 of each period, CSF samples will be collected at: 0 (pre-dose) and 1, 2, 4, 8, 12, 16, and 24 hours after dosing.

Safety assessments will include reporting of adverse events; clinical laboratory test results; vital sign measurements; electrocardiogram (ECG) results; and Columbia Suidical Severity Rating Scale (C-SSRS), Brief Psychiatric Rating Scale Positive Symptoms (BPRS+), and Clinician Administered Dissociative States Scale (CADSS) results. Adverse events, including serious adverse events (SAEs) and adverse events of special interest (AESIs), will be recorded from the time of informed consent until study completion.

ELIGIBILITY:
Inclusion Criteria:

* Available for the entire study period; willing and able to comply with the protocol requirements and study restrictions, to remain at the CRU for the required duration of the study, and to return for the Follow-Up Visit
* Male or female participants ≥18 to ≤59 years of age at Screening
* Minimum body weight of at least 50.0 kg at Screening
* Body mass index (BMI) 18.0 to 35.0 kg/m2, inclusive, at Screening
* Able and willing to swallow whole tablets without breaking, cutting, or chewing
* Non- or ex-smokers
* Considered generally healthy in the opinion of an investigator upon completion of medical history, physical examination, vital sign measurements, Screening clinical laboratory test results, and Screening ECG
* Female participants of childbearing potential must use an acceptable method of contraception, including hormonal contraceptives, abstinence from heterosexual intercourse, intrauterine device with or without hormones, or double-barrier method (eg, condom and spermicide) for 30 days before Screening, during the study, and for 30 days after the last administration of study drug
* Female participants of nonchildbearing potential should be surgically sterile (ie, have undergone complete hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or tubal ligation/occlusion) or in a menopausal state (at least 1 year without menses)
* Male participants must agree to use a double-barrier method (condom and spermicide) or remain abstinent from heterosexual intercourse at the time of Screening, during the study, and for 90 days after the last administration of study drug
* Male participants must agree not to donate sperm during the study and for 90 days after the last administration of study drug
* Able to fully consume the required fed meal within 30 minutes without substitutions
* Willing and able to provide written informed consent to participate in the study, is able to understand the procedures and study requirements, and agrees to comply with all required study requests and procedures
* Able to speak, read, and understand English sufficiently to allow completion of all study assessments

Exclusion Criteria:

* Female participant who is currently pregnant or lactating or is planning to become pregnant during the study
* Positive pregnancy test at Screening or on Day -1
* Positive test results for HIV 1/2 Ag/Ab, hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) at Screening
* Positive urine screen for drugs or alcohol at Screening or on Day -1
* Clinically significant history or evidence of gastrointestinal (excluding cholecystectomy), hepatic, renal, endocrine, pulmonary, neurologic, psychiatric, cardiovascular, hematologic, dermatologic, immunologic, or metabolic disease; or any other condition or organ system disease known to interfere with the absorption, distribution, metabolism, or elimination of drugs that in the opinion of an investigator would jeopardize the safety of the participant or impact validity of study results.
* Current or history of alcohol or substance abuse, with the exception of being fully recovered with no use of alcohol or substances of abuse within the 12 months before Screening
* Any clinically significant illness in the previous 30 days before Screening or Day -1
* Malignancy, a history of malignancy, or has received treatment for a malignancy at any time, with the exception of resected and cured basal cell carcinoma and squamous cell carcinoma of the skin (>1 year)
* Poor venous access
* Any medical condition(s) considered by an investigator to be clinically significant for study participation
* Supine pulse rate <60 or ≥100 bpm at Screening or on Day -1
* Donation or significant loss of blood products of 500 mL or more within 56 days before Screening, or donation or loss of plasma within 7 days before Screening
* Suicidal behavior or suicidal ideation of score 4 (active suicidal ideation with some intent to act without specific plan) or score 5 (active suicidal ideation with specific plan and intent) based on the C-SSRS within 12 months before Screening; a history of suicide attempt in the last 6 months; or more than 1 lifetime suicide attempt
* Positive responses on the CADSS or BPRS+ assessments at Screening, indicating evidence of dissociative symptoms or psychosis, as determined by the investigator
* Unable to abstain from consumption of grapefruit or Seville oranges or their juices from 14 days before the first administration of study drug until collection of the final PK sample
* Unable to abstain from caffeine- or xanthine-containing products (eg, coffee, tea, cola drinks, and chocolate) for 24 hours before admission to the clinical research unit until discharge
* Unable to abstain from alcohol for 48 hours before admission to the clinical research until discharge
* Unable to abstain from strenuous exercise for 48 hours before admission to the clincal research unit until after the collection of the final PK sample
* A marked prolongation of QT/corrected QT interval (QTc), defined as repeated QTc
* >450 ms for male participants and >470 ms for female participants using QT interval corrected for heart rate using Fridericia's formula (QTcF), at Screening or on Day -1
* Presence of observed abnormality (evidenced from physical examination, ECG [PR interval >220 ms, QRS >110 ms QRS or T wave morphology that in an investigator's opinion renders QT interval assessment unreliable], vital sign measurements, or clinical laboratory test results) considered by an investigator to be clinically significant for study participation. Out-of-range values can be repeated to confirm if the abnormality is sustained
* Use of any prescription medication (including oral contraceptives) within 14 days before Screening and/or use of any over-the-counter medications (such as antacids, vitamins, minerals, dietary/herbal preparations, and nutritional supplements) within 7 days before Screening
* Allergy to NMDA receptor drugs, to any component of the dosage form, or any other allergy, which, in the opinion of an investigator, contraindicates their participation
* Treatment with any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) before Screening
* Contraindications to lumbar puncture for CSF collection:
* Skin infection near the site of the lumbar puncture
* Significant scarring near the site (tattoos are acceptable)
* Uncorrected bleeding disorders
* Acute spinal cord trauma
* Suspicion of increased intracranial pressure due to a mass in the brain
* Significant degenerative changes or scoliosis of the lumbar spine
* Any reason that, in the opinion of the investigator, would prevent participation in the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameter Maximum Concentration (Cmax) in plasma | Hour zero to Hour 24
  Maximum concentration in plasma
Pharmacokinetic parameter Area Under the Curve (AUC) for Concentration in plasma over time | Hour 0 to hour 24
  Area under the curve from time 0 to hour 24
Pharmacokinetic parameter Maximum Concentration (Cmax) in cerebrospinal fluid | Hour 0 to Hour 24
  Maximum concentration in cerebrospinal fluid in plasma
Pharmacokinetic parameter Area Under the Curve (AUC) for concentration in cerebrospinal fluid over time | Hour 0 to hour 24
  Area under the curve from time 0 to hour 24 in cerebrospinal fluid

SECONDARY OUTCOMES:
Pharmacokinetic parameter Time of Maximum Concentration (Tmax) in plasma | Hour 0 to hour 24
  Time of maximum concentration in plasma
Pharmacokinetic parameter Elimination Half-Life (T1/2) in plasma | Hour 0 to hour 24
  Elimination half life in plasma
Pharmacokinetic parameter maximum concentration (Tmax) in cerebrospinal fluid | Hour 0 to hour 24
  Time of maximum concentration in cerebrospinal fluid
Pharmacokinetic parameter Elimination Half-Life (T1/2) in cerebrospinal fluid | Hour 0 to hour 24
  Ellimination half life in cerebrospinal fluid
Safety - Pulse Rate | Day -1 to Day 10
  Evaluation of pulse rate
Safety - Columbia Suicide Severity Rating Scale (C-SSRS) | Day -1 to day 10
  The C-SSRS assesses intensity of suicidal ideation with categories of increasing seriousness from Wish to be Dead (score 1), to Active Suicidal Ideation with Plan and Intent (score 5). The C-SSRS will be used to assess suicidal ideation and behaviors in participants who are able to complete the assessment.
Safety - Brief Psychiatric Rating Scale, positive symptoms (BPRS+) | Day -1 to Day 10
  Evaluation of changes in psychotic ideation in the areas of conceptual disorganization, suspiciousness, hallucinatory behavior, and unusual thought content, each of which is scored from 1 (normal) to 4 (severe) with increasing intensity for a total score from 4 to 16.
Safety - Clinician-Administered Dissociative States Scale (CADSS) | Day -1 to Day 10
  Evaluation of changes in dissociative symptoms in 23 areas, each of which is scored from 0 - not present to 4 - severe, for a total score from 0 to 92.
Safety - Treatment Emergent Adverse Events (TEAE) reported by subjects after treatment has begun | Day -1 to Day 10
  Evaluation of side effects experienced by subjects after drug treatment has begun
Safety Systolic Blood Pressure | Day -1 to Day 10
  Change in systolic blood pressure
Safety Diastolic Blood Pressure | Day -1 to Day 10
  Change in diastolic blood pressure
Safety Body Temperature | Day -1 to Day 10
  Change in body temperature
Safety Electrocardiogram QT Interval | Day -1 to Day 10
  Change in electrocardiogram QT interval
Safety Electrocardiogram PR Interval | Day -1 to Day 10
  Change in electrocardiogram PR interval
Safety Electrocardiogram QRS Interval | Day -1 to Day 10
  Change in electrocardiogram QRS interval
Pharmacodynamics EEG alpha power | Day -1 to Day 10
  Change in EEG alpha power
Safety estimated Glomerular Filtration Rate (eGFR) | Day -1 to Day 10
  Change in estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Burch Burch, MD, PhD, Study Director — Syndeio Biosciences, Inc
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No